CLINICAL TRIAL: NCT00730522
Title: Vigabatrin for Treatment of Methamphetamine Dependence: A Phase II Study
Brief Title: Safety and Efficacy Study of Vigabatrin to Treat Methamphetamine Dependence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: To conserve remaining capital, Sponsor decided to terminate the study early.
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPP-02001
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-10

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine; Dependency; Addiction; vigabatrin
MeSH Terms: conditions — Behavior, Addictive | interventions — Vigabatrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): CPP-109 vigabatrin tablets
  Interventions: Drug: CPP-109 vigabatrin
- 2 (Placebo Comparator): Matching Placebo Tablets
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: CPP-109 vigabatrin — tablets, bid for 12 weeks
  Other Names: GVG; gamma-vinyl GABA
  Arms: 1
Drug: Matching Placebo — tablets, bid, 12 weeks
  Arms: 2

SUMMARY:
The objective of this study is to demonstrate that a larger proportion of vigabatrin-treated subjects than placebo-treated subjects will be methamphetamine-free in the last 2 weeks of the study's Treatment Phase (Weeks 11 and 12).

DETAILED DESCRIPTION:
This is a Phase II, randomized, double-blind, placebo-controlled, intent-to-treat, 2-arm, parallel design, multicenter study to evaluate vigabatrin as a treatment for methamphetamine addiction. The study will involve approximately 180 subjects (90/group) who meet DSM IV criteria for methamphetamine dependence. Subjects will be evaluated for their compliance with protocol inclusion/exclusion criteria during Screening/Baseline Phase, lasting up to 4 weeks.

At the conclusion of the Screening/Baseline Phase, subjects meeting all inclusion/exclusion criteria will be randomized to one of two treatment groups: vigabatrin or placebo. Subjects will proceed to a 12 week Treatment Phase and then undergo a 12 week follow-up period. Subjects will be scheduled for clinic visits 3 times per week for efficacy and/or safety assessments during the Screening/Baseline Phase and the 12 week Treatment Phase. Subjects will return for follow up visits at Weeks 13, 16, 20 and 24.

ELIGIBILITY:
Inclusion Criteria:

Able to understand the study and provide written informed consent.

* Male or female at least 18 years of age.
* Meets DSM-IV (Diagnostic and Statistical Manual of Mental Disorders Fourth Edition) criteria for methamphetamine dependence as major diagnosis, as determined by the Substance Abuse module of SCID (Structured Clinical Interview for DSM-IV).
* Provides at least one urine specimen which is positive for methamphetamine according to a rapid screening test.
* Seeking treatment for methamphetamine dependence.
* Have normal visual fields.
* Be in generally good health based on history, physical examination and laboratory findings.
* If female of childbearing potential, use acceptable contraceptive methods

Exclusion Criteria:

* Has current dependence on any psychoactive substance other than methamphetamine, alcohol, nicotine, or cannabinoid or physiologic dependence on alcohol requiring medical detoxification.
* Has any serious medical or psychiatric illness and/or clinically significant abnormal laboratory values.
* Has history of serious cardiovascular reaction to methamphetamine.
* Has clinically significant cardiovascular impairment, abnormal ECG or uncontrolled hypertension.
* Be under court or other governmental agency (e.g. social services) mandate to obtain treatment or requiring outside urine monitoring.
* Be enrolled in an opiate substitution treatment program within 2 months of randomization.
* Has ever taken vigabatrin in the past.
* Is pregnant or lactating.
* Has clinically significant ophthalmologic disease, which would preclude safety monitoring, is undergoing treatment for ocular disease or intends to have any ocular surgery or procedure performed during the time of their participation in the trial.
* Has received a drug with known major organ toxicity, including retinotoxicity.
* Is currently participating in, or has been enrolled in another clinical trial within the last 30 days.
* Be anyone who, in the judgment of the investigator, would not be expected to attend regular study visits or to complete the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Gorodetzky, MD, PhD, Study Director — Catalyst Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - North County Clinical Research (NCCR), Oceanside, California
  - South Bay Treatment Center, San Diego, California
  - Addiction Pharmacology Research Laboratory, St. Luke's Hospital, San Francisco, California
  - START Research and Treatment, Kansas City, Missouri
  - Creighton University Medical Center, Omaha, Nebraska
  - Behavioral Health Research Center of the Southwest, Albuquerque, New Mexico
  - Pahl Pharmaceutical Research, Oklahoma City, Oklahoma
  - Pillar Research, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Vigabatrin Tablets: CPP-109 vigabatrin tablets (3.0 gm/day) for 12 weeks including 2 week dose escalation
  CPP-109 vigabatrin: tablets, bid for 12 weeks
- Matching Placebo Tablets: Matching Placebo Tablets for 12 weeks on a schedule to match active arm
  Matching Placebo: tablets, bid
Period: Overall Study
Arm/Group | Vigabatrin Tablets | Matching Placebo Tablets
Started | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated early due to failed trial in another category of substance dependence, very limited data summary performed and therefore most data not available, or not collected. What is available has been entered.
Groups:
- Vigabatrin: CPP-109 vigabatrin tablets
  CPP-109 vigabatrin: tablets, bid for 12 weeks
- Matching Placebo: Matching Placebo Tablets
  Matching Placebo: tablets, bid, 12 weeks
- Total: Total of all reporting groups
Arm/Group | Vigabatrin | Matching Placebo | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 44 [23 to 60] | 42 [26 to 54] | 43 [23 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 9 | 9 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55
Methamphetamine substance dependence [Count of Participants; unit: Participants] | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects in Each Treatment Group Who Are Amphetamine Abstinent During the Last 2 Weeks of the Treatment Phase (Weeks 11 and 12).
Time Frame: Weeks 11-12
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Matching Placebo Tablets
  Matching Placebo: tablets, bid, 12 weeks
Arm/Group | Vigabatrin | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 4 | 2

2. Secondary Outcome: • Number of Methamphetamine Negative Urines During the Treatment Phase • Number of Methamphetamine Use Weeks During the Treatment Phase.
Time Frame: Weeks 1-12
Population: Data were not collected due to early study termination.
Groups:
- CPP-109 Vigabatrin Treated Group: Participants who received CPP-109 (vigabatrin) tablets
  CPP-109 vigabatrin: tablets, bid for 12 weeks
- Matching Placebo Treated Group: Participants who received Matching Placebo Tablets
  Matching Placebo: tablets, bid, 12 weeks
Arm/Group | CPP-109 Vigabatrin Treated Group | Matching Placebo Treated Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Vigabatrin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/28 | 0/27
Other Adverse Events (participants affected / at risk) | 24/28 | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vigabatrin (N=28) | Placebo (N=27)
Hernia obstructive (General disorders) | 1 | 0 — Subject had an incisional hernia on the anterior abdominal wall prior to study, which became incarcerated and required surgical repair.
fracture (Injury, poisoning and procedural complications) | 1 | 0 — Subject fell off of a ladder and broke left arm.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vigabatrin (N=28) | Placebo (N=27)
Fatigue (General disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 2
Depression (Psychiatric disorders) | 0 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Somnolence (Psychiatric disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 3
Tooth infection (Infections and infestations) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Ovarian Cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study terminated early due to other failed indication for product and only limited data collected without complete analysis. CPP-109 stopped all development in substance dependent indications. Therefore, not able to summarize most data, as not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No